CLINICAL TRIAL: NCT02324842
Title: Effect of Combined Incretin-Based Therapy Plus Canagliflozin on Glycemic Control and the Compensatory Rise in Hepatic Glucose Production in Type 2 Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 28431754DIA4009; HSC20140322H (Other: University of Texas Health Science Center- San Antonio)
Record Dates: First submitted 2014-11-10; First posted 2014-12-24 (Estimated); Results first posted 2019-05-14 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Canagliflozin; Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Canagliflozin (Active Comparator): canagliflozin (film-coated tablet), 100 mg/day, increased to 300 mg/day after week two if tolerated without side effects
  Interventions: Drug: Canagliflozin
- liraglutide (Active Comparator): liraglutide, 1.2 mg/day, increased to 1.8 mg/day after week two if tolerated without side effects
  Interventions: Drug: Liraglutide
- canagliflozin plus liraglutide (Active Comparator): canagliflozin, 100 mg/day, plus liraglutide, 1.2 mg/day, increased to 300 mg/day and 1.8 mg/day, respectively at week two, if tolerated without side effects
  Interventions: Drug: Canagliflozin; Drug: Liraglutide

INTERVENTIONS:
Drug: Canagliflozin — Canagliflozin is a sodium-glucose co-transporter 2 (SGLT2) inhibitor indicated as an adjunct to diet and exercise to improve glycemic control in adults with type 2 diabetes mellitus (1)
  Other Names: Invokana
  Arms: Canagliflozin; canagliflozin plus liraglutide
Drug: Liraglutide — Liraglutide is a glucagon-like peptide-1 (GLP-1) receptor agonist indicated as an adjunct to diet and exercise to improve glycemic control in adults with type 2 diabetes mellitus.
  Other Names: Victoza
  Arms: canagliflozin plus liraglutide; liraglutide

SUMMARY:
Specific Aim 1.To examine whether the combination of liraglutide plus canagliflozin can prevent the increase in Hepatic Glucose Production (HGP) following institution of canagliflozin therapy and produce an additive or even synergistic effect to lower the plasma glucose concentration and A1c.

Specific Aim 2: To examine whether combination therapy with liraglutide plus canagliflozin can produce an additive, or even synergistic, effect to promote weight loss and reduction in hepatic and visceral fat content.

Specific Aim 3. To examine whether combination therapy with liraglutide plus canagliflozin can produce an additive or even synergistic effect to reduce systolic/diastolic blood pressure and 24-hour integrated blood pressure.

DETAILED DESCRIPTION:
Specific Aim 1.To examine whether the combination of liraglutide plus canagliflozin can prevent the increase in HGP following institution of canagliflozin therapy and produce an additive or even synergistic effect to lower the plasma glucose concentration and A1c. We will examine this hypothesis by comparing the effect of administration of liraglutide alone, canagliflozin alone, and the combination of liraglutide plus canagliflozin on:(i) the rate of HGP; (ii) decrease in fasting plasma glucose concentration; (iii) counter-regulatory hormone response and (iv) A1c. We anticipate that the addition of liraglutide to canagliflozin will prevent the increase in plasma glucagon concentration, augment insulin secretion, and blunt/block the increase in HGP in response to canagliflozin, resulting in a greater decrease in fasting plasma glucose concentration and A1c than observed with each therapy alone.

Specific Aim 2: To examine whether combination therapy with liraglutide plus canagliflozin can produce an additive, or even synergistic, effect to promote weight loss and reduction in hepatic and visceral fat content.

Specific Aim 3. To examine whether combination therapy with liraglutide plus canagliflozin can produce an additive or even synergistic effect to reduce systolic/diastolic blood pressure and 24-hour integrated blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between the ages of 18-70
* Subjects with Type 2 Diabetes Mellitus (T2DM)
* Drug naïve or on stable dose (more than 3 months) of metformin with or without sulfonylurea
* Have an HbA1c levels ≥7.0% and <10.0%
* Stable weight (± 3 lbs) over the preceding 3 months

Exclusion Criteria:

* Subjects taking drugs known to affect glucose metabolism (other than metformin) will be excluded.
* Individuals with evidence of proliferative diabetic retinopathy or plasma creatinine >1.4 females or >1.5 males or estimated Glomerular Filtration Rate (eGFR)< 60 ml/min.172m2 will be excluded
* Unstable body weight (change of greater than ±3 lbs over the preceding 3 months)
* Participates in excessively heavy exercise program

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-11; Primary Completion 2018-03-28 (Actual); Study Completion 2019-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugenio Cersosimo, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

REFERENCES:
- [Derived] Ali AM, Mari A, Martinez R, Al-Jobori H, Adams J, Triplitt C, DeFronzo R, Cersosimo E, Abdul-Ghani M. Improved Beta Cell Glucose Sensitivity Plays Predominant Role in the Decrease in HbA1c with Cana and Lira in T2DM. J Clin Endocrinol Metab. 2020 Oct 1;105(10):dgaa494. doi: 10.1210/clinem/dgaa494. PMID 32745202
- [Derived] Ali AM, Martinez R, Al-Jobori H, Adams J, Triplitt C, DeFronzo R, Cersosimo E, Abdul-Ghani M. Combination Therapy With Canagliflozin Plus Liraglutide Exerts Additive Effect on Weight Loss, but Not on HbA1c, in Patients With Type 2 Diabetes. Diabetes Care. 2020 Jun;43(6):1234-1241. doi: 10.2337/dc18-2460. Epub 2020 Mar 27. PMID 32220916

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Canagliflozin | Liraglutide | Canagliflozin Plus Liraglutide
Started | 15 | 15 | 15
Completed | 14 | 14 | 13
Not Completed | 1 | 1 | 2
Not completed — Lost to Follow-up | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Canagliflozin | Liraglutide | Canagliflozin Plus Liraglutide | Total
Number analyzed (Participants) | 14 | 14 | 13 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 13 | 41
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 7 | 17
  Male | 10 | 8 | 6 | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 13 | 41

OUTCOME MEASURES:

1. Primary Outcome: HbA1c at 4 Months
Description: Primary end point of the study is the HbA1c level in response to canagliflozin alone, liraglutide or canagliflozin with liraglutide.
Time Frame: Approximately 4 months
Measure: Mean (Standard Deviation); unit: percentage glycated hemoglobin
Arm/Group | Canagliflozin | Liraglutide | Canagliflozin Plus Liraglutide
Number analyzed (Participants) | 15 | 15 | 15
percentage glycated hemoglobin | 8.2 (0.3) | 8.4 (0.3) | 8.1 (0.3)

2. Primary Outcome: Fasting Plasma Glucose (FPG) at 4 Months
Description: Values will be presented as the mean + (Standard Deviation) SD. The difference in HGP and all secondary endpoints at study end versus baseline will be calculated and compared between each active treatment group with ANOVA.
Time Frame: Baseline to Approximately 4 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Canagliflozin | Liraglutide | Canagliflozin Plus Liraglutide
Number analyzed (Participants) | 15 | 15 | 15
mg/dl | 174 (12) | 177 (10) | 180 (15)

3. Secondary Outcome: Body Mass Index (BMI) at 4 Months
Description: A measure of BMI at 4 months to examine effects of combination therapy with liraglutide plus canagliflozin.
Time Frame: Approximately 4 months
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Canagliflozin | Liraglutide | Canagliflozin Plus Liraglutide
Number analyzed (Participants) | 15 | 15 | 15
kg/m2 | 34.8 (1.7) | 35.1 (1.1) | 34.8 (1.1)

4. Other Pre Specified Outcome: Change in Matsuda Index of Insulin Sensitivity, Insulin Secretion, and Beta Cell Function During Oral Glucose Tolerance Test (OGTT)
Description: Values will be presented as the mean + SD. The Matsuda Index is a novel assessment of insulin sensitivity that is simple to calculate and provides a reasonable approximation of whole-body insulin sensitivity from the OGTT. The index is calculated from plasma glucose (mg/dl) and insulin (mIU/l) concentrations in both fasting state and post-OGTT. The index value obtained is compared to normal physiologic values to assess insulin sensitivity or resistance. The higher the number, the more insulin sensitive and the lower the number the more insulin resistant the subjects are. Insulin secretion will be measured from plasma C-peptide concentration during the OGTT and the Mari Model will be used to measure beta cell glucose sensitivity
Time Frame: Change from Baseline to Approximately 4 months
Measure: Mean (Standard Deviation); unit: index value
Arm/Group | Canagliflozin | Liraglutide | Canagliflozin Plus Liraglutide
Number analyzed (Participants) | 15 | 15 | 15
index value | 0.8 (0.4) | -0.5 (0.4) | 0.1 (0.2)

5. Other Pre Specified Outcome: Change in Free Plasma Insulin at the End of the Study From Baseline Value
Description: Values will be presented as the mean + SD. The difference in HGP and all secondary endpoints at study end versus baseline will be calculated and compared between each active treatment group with ANOVA.
Time Frame: At Approximately 4 months
Measure: Mean (Standard Deviation); unit: mg/ml
Arm/Group | Canagliflozin | Liraglutide | Canagliflozin Plus Liraglutide
Number analyzed (Participants) | 15 | 15 | 15
mg/ml | -2 (2) | 2 (2) | 0.7 (1)

6. Other Pre Specified Outcome: Change in Plasma Glucagon Concentration at the End of the Study Compared to Baseline
Description: as for outcome 5
Time Frame: Approximately 4 months
Measure: Mean (Standard Deviation); unit: mg/ml
Arm/Group | Canagliflozin | Liraglutide | Canagliflozin Plus Liraglutide
Number analyzed (Participants) | 15 | 15 | 15
mg/ml | 12 (6) | -7 (5) | -5 (5)

7. Other Pre Specified Outcome: Change in Total Body Weight at Study End Compared to Baseline
Description: Values will be presented as the mean + SD. The difference in HGP and all secondary endpoints at study end versus baseline will be calculated and compared between each active treatment group with ANOVA. The difference between baseline and study end will represent the change in body weight due to change in hepatic, visceral and abdominal subcutaneous fat.
Time Frame: Approximately 4 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Canagliflozin | Liraglutide | Canagliflozin Plus Liraglutide
Number analyzed (Participants) | 15 | 15 | 15
kg | -3.5 (0.5) | -1.9 (.8) | -6.0 (0.8)

8. Other Pre Specified Outcome: Change in 24-hour Blood Pressure at Study End Compared to Baseline.
Description: as for outcome 5
Time Frame: Approximately 4 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Canagliflozin | Liraglutide | Canagliflozin Plus Liraglutide
Number analyzed (Participants) | 15 | 15 | 15
mmHg | -5.2 (2.2) | 5.1 (3.8) | -14.1 (3.0)

ADVERSE EVENTS:
Time Frame: Adverse Events were reported from Baseline to 4 months
Arm/Group | Canagliflozin | Liraglutide | Canagliflozin Plus Liraglutide
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 13/15 | 13/15 | 12/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Canagliflozin (N=15) | Liraglutide (N=15) | Canagliflozin Plus Liraglutide (N=15)
Dehydration/Hyperkalemia (General disorders) | 1 (1) | 0 (0) | 0 (0) — Subject was hospitalized and dehydration and hyperkalemia resolved
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Canagliflozin (N=15) | Liraglutide (N=15) | Canagliflozin Plus Liraglutide (N=15)
Nausea (Gastrointestinal disorders) | 1 (1) | 9 (11) | 8 (12)
Dry Mouth (Gastrointestinal disorders) | 4 (5) | 0 (0) | 6 (7)
Abdominal Discomfort (Gastrointestinal disorders) | 3 (3) | 7 (11) | 4 (4)
Decreased Appetite (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2)
Gastrointestinal Reflux/Indigestion (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (7)
Constipation (Gastrointestinal disorders) | 0 (0) | 5 (5) | 5 (6)
Urinary Frequency increased (Renal and urinary disorders) | 13 (15) | 0 (0) | 3 (3)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Light-headedness/Dizziness (Nervous system disorders) | 4 (5) | 1 (1) | 2 (3)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Anxiety (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (3) | 2 (2) | 1 (1)
Redness at Injection Site (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bilateral Leg Cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Cough and nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Symptomatic Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 3 (3)
Vaginal Candidiasis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 3 (3)
Vaginal itching or foreskin pain (Reproductive system and breast disorders) | 2 (3) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-19): https://cdn.clinicaltrials.gov/large-docs/42/NCT02324842/Prot_SAP_000.pdf